CLINICAL TRIAL: NCT01765842
Title: Comparison of the Efficacy of Two Rituximab Treatment Regimens in Patients With Lupus Nephropathy Resistant to Conventional Treatments.
Brief Title: Comparison of the Efficacy of Two Rituximab Treatment Regimens in Patients With Lupus Nephropathy
Acronym: RITULUP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The recruitment period has finished without reaching sample size
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RITULUP
Record Dates: First submitted 2013-01-03; First posted 2013-01-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2013-01

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; remission; immunosuppressive treatment
MeSH Terms: conditions — Lupus Nephritis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab (1 cycle) (Active Comparator): 1 cycle of Rituximab (4 i.v. infusions):
  Day 0: 375 mg/m2 Day 7: 375 mg/m2 Day 14: 375 mg/m2 Day 21: 375 mg/m2
  Interventions: Biological: Rituximab
- Rituximab (2 cycles) (Experimental): A second cycle of Rituximab
  First cycle of Rituximab (4 i.v. infusions):
  Day 0: 375 mg/m2 Day 7: 375 mg/m2 Day 14: 375 mg/m2 Day 21: 375 mg/m2
  Second cycle of Rituximab (4 i.v. infusions, 6 months later)
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: Rituximab — Only one cycle of rituximab will be administered in this arm.
  Other Names: Mabthera

SUMMARY:
Comparison of the Efficacy of Two Rituximab Treatment Regimens in Patients With Lupus Nephropathy Resistant to Conventional Treatments

DETAILED DESCRIPTION:
Randomized, open, controlled, multicenter, clinical trial in patients with lupus nephritis previously treated with cyclophosphamide and mycophenolate. These patient can not have received Rituximab in the previous year. The number of patients estimated to reach statistical significance is 18 in each arm, a total sample size of 32 patients is needed.

The hypothesis is that the alternative procedure (a second cycle of Rituximab)will reduce the relapse rate of lupus nephritis and the consequent deterioration of renal function. Besides it will reduce health care expenses(hospitalization, medication, hemodialysis and renal transplantation).

ELIGIBILITY:
Inclusion Criteria:

* Both men and women between 18 and 70 years.
* Patient with active lupus nephritis, previously treated with cyclophosphamide and mycophenolate (sodium or mofetil), who have not received rituximab in the previous year.
* Women in childbearing age must have a pregnancy test in serum or urine negative and should use a contraceptive method suitable since at least 14 days prior to their inclusion in the study and up to 6 months after the last dose of the medication of the test.
* Informed consent form signed.

Exclusion Criteria:

* Patients treated with rituximab in the previous years
* Active/sepsis serious infections
* Renal biopsy showing interstitial fibrosis and/or glomerular over 75%.
* Known neoplasia
* Heart failure with III/IV functional class
* Pregnancy
* Nursing
* Known anaphylaxis to the product
* History of hepatitis c
* History of tuberculosis
* Cardiovascular disease or uncontrolled hypertension
* Chronic hepatitis B
* Serious Cytopenia (granulocytes < 500/mm3, further < 10000/mm3)
* Immunodeficiency (CVI, immunoglobulins deficiency)
* Infection with HIV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Rate of complete or partial response in lupus nephritis | Assessment at 12 months
  Complete response defined as:
  * Glomerular Filtration Rate (GFR)≥ 60, 73 m2 (or decline to baseline or
    ± 15% of baseline in those with GFR <60 ml/min/1, 73m2).
  * Proteinuria ≤ 0.5 g/24 hours.
  * Inactive urine sediment (red cells, white cells, red cell casts according to local laboratory ranges).
  * Serum albumin> 3 g / dl
  Partial response defined as:
  In patients with proteinuria ≥ 3.5 gr/24 h , decreased proteinuria <3.5 gr/24 hours.
  * In patients with baseline proteinuria <3.5 gr/24 hours, reduced proteinuria> 50% of baseline.
  * In both situations, stabilization (± 25%) or reduce of the Glomerular Filtration Rate.

SECONDARY OUTCOMES:
Renal function | 24 months of follow-up
  Proportion of patients achieving a stabilization of renal function (Glomerular filtration rate of ± 25% over baseline or serum creatinine within normal range)
Safety | 24 months of follow-up
  Incidence of adverse events, serious adverse events and adverse events that led to the interruption of the study.
Rescue medication | 24 months of follow-up
  Need for immunosuppressive treatment added to the experimental pattern:
  1. - Mycophenolate
  2. - Azathioprine
  3. - Methotrexate
Efficacy | 24 months of follow-up
  Improvements in Selena-SLEDAI (Systemic Lupus Erythematosus Disease Activity Index) score results

CONTACTS AND LOCATIONS:
Overall Officials: María Jesús Castillo Palma, PhD, Study Chair — Virgen del Rocío Hospital
Locations (3):
- Spain (3):
  - San Cecilio Hospital, Granada, Granada
  - Carlos Haya Hospital, Málaga, Málaga
  - Virgen del Rocío, Hospital, Seville, Seville